CLINICAL TRIAL: NCT01923064
Title: A Randomized Study to Compare Effect of Endoscopic Injection of a Mixture of Cyanoacrylate and Lipiodol Versus Cyanoacrylate and Lauromacrogol in Gastric Varices
Brief Title: Injection of Cyanoacrylate+Lipiodol vs Cyanoacrylate+Lauromacrogol in Gastric Varices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: chen2013
Record Dates: First submitted 2013-08-07; First posted 2013-08-14 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Gastric Varices; Portal Hypertension
MeSH Terms: conditions — Esophageal and Gastric Varices; Hypertension, Portal | interventions — Ethiodized Oil; Polidocanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NBCA-lipiodol (Active Comparator): Patients will receive injection of a mixture of cyanoacrylate and lipiodol to treat gastric varices
  Interventions: Drug: Lipiodol
- NBCA-lauromacrogol (Experimental): Patients will receive injection of the mixture of cyanoacrylate and lauromacrogol to treat gastric varices
  Interventions: Drug: Lauromacrogol

INTERVENTIONS:
Drug: Lipiodol — endoscopic injection of lipiodol + cyanoacrylate + lipiodol for gastric varices
  Arms: NBCA-lipiodol
Drug: Lauromacrogol — endoscopic injection of lauromacrogol + cyanoacrylate + lauromacrogol for gastric varices
  Arms: NBCA-lauromacrogol

SUMMARY:
The purpose of this randomized study to compare effect of endoscopic injection of a mixture of cyanoacrylate and lipiodol versus cyanoacrylate and lauromacrogol in gastric varices.

DETAILED DESCRIPTION:
Gastroesophageal variceal bleeding is known as one of the most frequent death causes of patients with portal hypertension. When a patient has a bleeding episode, if no further prophylactic treatments is given, it's very likely that he/she will develop another rebleeding event in the future and maybe a terminal event. Gastric varices occur in 18-70% of patients with portal hypertension, which appear to be more severe, to require more transfusion and to have a higher mortality rate than esophageal variceal bleeding, with a high rate of rebleeding(38-89%). It has been recommended to use endoscopic cyanoacrylate injection as the first line treatment for hemostasis and secondary prophylaxis for gastric varices by general consensus. However, the efficacy and prevalence of complications between mixture of cyanoacrylate + lipiodol and cyanoacrylate + lauromacrogol have not yet been explored and reported. We conducted this study to evaluate the effect of endoscopic injection of a mixture of cyanoacrylate and lipiodol versus cyanoacrylate and lauromacrogol in gastric varices.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented to our hospital with acute gastric variceal bleeding, with or without liver cirrhosis.
* The age of the patients range from 18 to 80 years old.

Exclusion Criteria:

* Patients who have contraindications for cyanoacrylate, lipiodol or lauromacrogol therapy.
* Patients who have abnormal portosystemic shunt according to the imaging results.
* Patients who have no previous upper gastrointestinal bleeding history.
* Patients who have multiple endoscopic treatments for esophagogastric varices before.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
bleeding rate of the puncture site | time period since the beginning of the injection, until up to 24 hours after the procedure
  We tend to observe the immediate puncture site bleed on the injection of cyanoacrylate and lipiodol or lauromacrogol and withdrawal of needle catheter during endoscopic treatment of gastric varices.

SECONDARY OUTCOMES:
Rebleeding rate after endoscopic treatment | 6 months from the date of enrollment
  Patients were followed up for 6 months to see if they experience relapse of bleeding, presenting melena, haematemesis or both.

OTHER OUTCOMES:
incidence rate of ulcer formation | 2 months after the initial endoscopic treatment
  The patients will be assessed if ulceration is formed on the site of the injection when they have gastroscopy review in 2 months after the initial endoscopic treatment.
eradication rate of gastric varices | 2 months after the initial endoscopic treatment
  Patients will be evaluated if gastric varices are eradicated when they have gastroscopy review in 2 months after the initial endoscopic treatment.
incidence rate of complications | 6 months
  Participants will be followed for up to 6 months starting from the date of enrollment.Complications associated with endoscopic treatments include transient fever, transient dysphagia, transient arrhythmias, ulceration, perforation, stricture, rebleeding, aspiration pneumonia, sepsis, peritonitis and chest pain.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, MD, Study Director — Zhongshan Hospital, Shanghai
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China